CLINICAL TRIAL: NCT05510440
Title: Effect of Supplementation With Alpha-amino Acid Derivatives on the Level of Systemic Inflammatory Response and Post-workout Kidney Damage in Long Distance Runners
Brief Title: Supplementation With Altha-aminoacids and Systemiec Inflammatory Response in Long-distance Runners.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MUGdansk Citrulline
Record Dates: First submitted 2022-06-20; First posted 2022-08-22 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Exercise Myoglobinuria; Citrulline; Metabolic Disorder; Iron Metabolism Disorders; Inflammatory Response
MeSH Terms: conditions — Metabolic Diseases; Iron Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of citrulline supplementation combined with long distance running on systemic inflammation (Experimental): 14-day protocol of supplementation with 6 g of citrulline.
  Interventions: Dietary Supplement: Alpha-amino acid derivatives
- Effect of placebo supplementation combined with long distance running on systemic inflammation (Placebo Comparator): 14-day protocol of supplementation with 6 g of placebo.
  Interventions: Dietary Supplement: Alpha-amino acid derivatives

INTERVENTIONS:
Dietary Supplement: Alpha-amino acid derivatives — Alpha-amino acid derivatives mainly citrulline will be used as a supplement to reduce kidneys and other internal organs damage

SUMMARY:
It is also noteworthy that the imbalance between the production, supply and elimination of especially α-amino acids may contribute to the intensification of the inflammatory response and the subsequent burden of the renal tubules, which may result in damage and developing chronic renal failure.

Among the many amino acids used in sports, arginine and its metabolites deserve special attention. The role of arginine appears to increase in specific physiological states associated with disease, injury or significant strain on the body, leading to an increase in the rate of catabolic transformation.

Arginine plays a significant role in protein biosynthesis and detoxification processes related to ammonia removal and urea formation .

DETAILED DESCRIPTION:
Subject and purpose of the project. Both in sport and medicine, methods are constantly being sought that can significantly contribute to improving the ability of tissues to perform their functions. A wide range of interests include various supplementation and training protocols. In a significant way, they are to contribute to the reduction of negative post-workout changes, protecting the athlete's tissues and organs from the debilitating effect of efforts of very long duration and high intensity.

Commonly, in sports with a long duration of effort, supplementation with amino acid complexes is used, the purpose of which is to support both the metabolism of working muscles and provide building materials necessary for the functioning of muscle fibers. It was found that maintaining a proper supply of amino acids is one of the important factors protecting the human body against excessive intensification of catabolic processes.

It is also noteworthy that the imbalance between the production, supply and elimination of especially α-amino acids may contribute to the intensification of the inflammatory response and the subsequent burden of the renal tubules, which may result in damage and developing chronic renal failure.

Among the many amino acids used in sports, arginine and its metabolites deserve special attention. The role of arginine appears to increase in specific physiological states associated with disease, injury or significant strain on the body, leading to an increase in the rate of catabolic transformation Arginine plays a significant role in protein biosynthesis and detoxification processes related to ammonia removal and urea formation In addition, it was found that arginine is involved in the synthesis of proline, and may have a special effect on the body of athletes: creatine, nitric oxide, agmatine, ornithine, citrulline and glutamate. Attention is also drawn to the possible relationship between arginine and the secretion of endogenous growth hormone, insulin and glucagon . It is noteworthy that as a result of digestion, only 50% of arginine consumed with the diet after its release from proteins enters the blood, while 40% is broken down in the small intestine as a result of arginase . Part of the arginine pool in the blood plasma may come from the conversion of citrulline found in food.

In cells, arginine transport takes place via specific membrane conveyors and is competently inhibited by selected NOS inhibitors (nitric oxide synthesis) and lysine, ornithine and canvaaine. In the liver, it participates in important detoxification processes, taking part in the urea cycle, while in vascular endothelial cells it stimulates the synthesis of nitric oxide.

The dietary supply of arginine, unfortunately, is not effective. A much greater increase in its content in blood plasma is observed in the case of the use of an increased arginine precursor - citrulline.

This means that thanks to the correct content of citrulline in the diet, it is possible to normalize the concentration of arginine in the body.

In the case of physical activity itself, however, it seems more important that the high supply of citrulline in the diet may translate into an increase in oxygen consumption by tissues, improvement of strength capabilities, but what is very important, it may have a positive effect on bicarbonate reuptake, which is an exponent of normal kidney function. In addition, by limiting muscle damage and the breakdown of muscle fibers, the myoglobin content in the urine is reduced. In turn, its high concentration (>35 ng / ml or above 17 μg / g creatinine) is considered an important factor responsible for post-workout kidney damage.

Suplementacjand citrulline in the case of ultramarathoners in terms of kidney function seems to be a very beneficial solution. The transformation of citrulline into arginine may translate into an increase in the concentration of nitrous oxide in the musculature of the renal vessels, which reduces the risk of ischemic changes developing in the kidney structure itself.

Summing up the above properties of citrulline and the achievable benefits of its use, the subject of a smaller research project is to determine the effect of citrulline supplementation on the level of generalized inflammatory reaction induced by ultralong physical exertion.

The aim of the entire research project is to try to show the phenomenon of post-workout kidney damage occurring in ultralong runners, as well as to illustrate the need to take (supplementation) actions aimed at protecting the kidneys, especially against toxic imbalance in the turnover of amino acids and the intensification of the harmful inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Men over 21 years of age with good health confirmed in a medical examination,
* training long runs with a confirmed minimum of five participation and completion of ultra-long runs (>42km)

Exclusion Criteria:

* neuromuscular diseases,
* cardiovascular disorders,
* cancer,
* hyperparathyroidism and thyroid,
* dementia disorders and other diseases of the nervous and circulatory systems that may significantly contribute to problems with the implementation of research tasks

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Systemic inflammation | 14 days
  Determining whether the 14-day protocol of supplementation with 6 g of citrulline contributes to the reduction of the inflammatory response, concentration of serum proinflammatory cytokines will be measured by multiplex technique
Post workout kidney damage , | 14 days
  Determining whether the 14-day protocol of supplementation with 6 g of citrulline contributes to kidney damage induced by running, concentration of serum and urine markers of kidney function will be measured by standard methods.
Internal organe damage | 14 days
  Determining whether the 14-day protocol of supplementation with 6 g of citrulline contributes to the reduction internal organs damage induced by running effort, concentration of serum markers of heart, liver, and kidney and skeletal muscle damage will be measured by multiplex technique.

CONTACTS AND LOCATIONS:
Overall Officials: Jędrzej Antosiewicz, Principal Investigator — Medical University of Gdańsk, Poland
Locations (2):
- Poland (2):
  - Medical University of Gdańsk Faculty of Health Science, Gdansk, Pomeranian Voivodeship
  - Medical University of Gdańsk, Gdansk

IPD SHARING:
Plan to Share IPD: Yes
Under reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: for two years after the publication of the results
Access Criteria: Reasonable request